CLINICAL TRIAL: NCT05715060
Title: Stainless Steel Wire vs. Polydioxanone "PDS" at Sternal Closure in Children After Cardiac Surgery
Brief Title: Sternal Closure in Children After Cardiac Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mostafa Ibrahim Mohammad AbdelHafeez, Resident, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: sternal closure in children
Record Dates: First submitted 2022-11-08; First posted 2023-02-06 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Open Heart Surgery

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- stainless steel wire closure (Active Comparator): conventional closure of median sternotomy by stainless steel wire
  Interventions: Procedure: Median sternotomy closure (sternal closure)
- PDS sternal closure (Active Comparator): closure of median sternotomy by PDS
  Interventions: Procedure: Median sternotomy closure (sternal closure)

INTERVENTIONS:
Procedure: Median sternotomy closure (sternal closure) — Comparison of Sternal closure after cardiac surgery between conventional way which is by stainless steel wire & Polydioxanone (PDS)

SUMMARY:
comparison between stainless steel wires and PDS in closure of sternum in children after cardiac surgery in terms of sternal dehiscence, infection & cosmetic outcome

DETAILED DESCRIPTION:
Median sternotomy is considered to be the gold standard incision in cardiac surgery. Sternotomy has to be performed properly to avoid short- and long-term morbidity and mortality. The surgical technique is well established and certain principles are recognized to be crucial to minimize complications. The identification of the correct landmarks, midline tissue preparation, osteotomy with the avoidance of injury to underlying structures like pleura, pericardium and ectatic ascending aorta, and targeted bleeding control are important steps of the procedure. As important as the performance of a proper sternotomy is a correct sternal closure. An override or shift of the sternal edges has to be avoided by placing the wires at a proper distance from each other without injuring the thoracic pedicle. The two sternal halves have to be tightly re-approximated to facilitate healing of the bone and to avoid instability, which is a risk factor for wound infection. With a proper performance of sternotomy and sternal closure, instability and wound infections are rare and depend on patient-related risk factors . Conventional closure uses stainless steel wire sutures which may not be the ideal approach as sternal wound infection and mediastinitis are troublesome complications following this method which are major causes of morbidity and mortality of patients. Availability of delayed absorbable sutures such as polydioxanone sutures (PDS) for sternal closure allows us to test the efficacy of it in prevention of these complications.

ELIGIBILITY:
Inclusion Criteria:

* Infants & children up to 5 years old underwent open heart surgery in Assiut University heart hospital

Exclusion Criteria:

* Older than 5 years old

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Sternal stability | up to 2 years
  Comparison of incidence of sternal dehiscence & instability between 2 groups this is done by clinical assessment(history & examination) & follow up chest x-rays

SECONDARY OUTCOMES:
cosmetic outcome (prominent wire) | up to 2 years
  calculation and observation of prominent wire incidence in patients closed with stainless steel wire Done by clinical assessment(history & examination)
Wound infection | up to 2 years
  comparison of incidence of skin infection between 2 groups Done by clinical assessment(history & examination)

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University heart hospital, Asyut, Egypt